CLINICAL TRIAL: NCT03732118
Title: EYE-Mobile TRACKer IN the Diagnosis of Minimal Hepatic Encephalopathy
Acronym: EyeMTRACKIN-HE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17058J; 2018-A02156-49 (Other: ANSM)
Record Dates: First submitted 2018-10-22; First posted 2018-11-06 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-02

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimal hepatic encephalopathy
  Interventions: Device: Eye-tracker Mobile EBT
- No hepatic encephalopathy (minimal or clinical)
  Interventions: Device: Eye-tracker Mobile EBT

INTERVENTIONS:
Device: Eye-tracker Mobile EBT — Use of the eye-tracker for the diagnosis of minimal HE by studying the characteristics of saccades and anti-saccades during a day hospitalization.

SUMMARY:
Hepatic encephalopathy (HE) corresponds to the neurological or the neuropsychological symptoms caused by an acute or chronic liver disease and/or porto-systemic shunt. Many patients present neurological symptoms even if their liver disease is stabilized. Furthermore, HE is associated with an altered quality of life and an increased mortality. Its incidence is high with 30 to 80% of cirrhotic patients that will display according to retained diagnostic criteria. HE symptoms are going from subtle neuropsychological abnormalities detected only on neuropsychological testing, minimal HE, to altered consciousness, overt HE. Recently, the therapeutic armamentarium has increased with now several drugs (rifaximin, ammonia lowering agents) that are able to prevent new bouts of HE. Unfortunately, the diagnosis of minimal HE is difficult and no gold-standard is available. None of the proposed test is rapid and easily performed at bedside.

Recently, different studies suggest the potential interest of the study of the ocular movements in HE. Abnormalities in ocular saccades could be an early predictor of cortical impairment. In a pilot feasibility study using an eye-tracker, we could show that cirrhotic patients with minimal HE had, compared to healthy controls, increased latencies, decreased speed of voluntary and reflex saccades, more errors in anti-saccades, more anticipations saccades and more difficulties to fix the target.

Our hypothesis was that the use of the eye-tracker will enable the diagnosis of minimal HE by studying the characteristics of saccades and anti-saccades.

Since no gold-standard is available for the diagnosis of minimal HE, we will use the conclusion of an adjudication committee formed by 2 experts. Their clinical judgment will take into account the results of medical history, clinical examination, neuropsychological testing, PHES, Critical Flicker Frequency test (CFF), ammonemia levels, EEG and brain MRI with spectroscopy.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) corresponds to the neurological or the neuropsychological symptoms caused by an acute or chronic liver disease and/or porto-systemic shunt. Many patients present neurological symptoms even if their liver disease is stabilized. Furthermore, HE is associated with an altered quality of life and an increased mortality. Its incidence is high with 30 to 80% of cirrhotic patients that will display according to retained diagnostic criteria. HE symptoms are going from subtle neuropsychological abnormalities detected only on neuropsychological testing, minimal HE, to altered consciousness, overt HE. Recently, the therapeutic armamentarium has increased with now several drugs (rifaximine, ammonia lowering agents) that are able to prevent new bouts of HE. Unfortunately, the diagnosis of minimal HE is difficult and no gold-standard is available. None of the proposed test is rapid and easily performed at bedside.

Recently, different studies suggest the potential interest of the study of the ocular movements in HE. Abnormalities in ocular saccads could be an early predictor of cortical impairment. In a pilot feasibility study using an eye-tracker, we could show that cirrhotic patients with minimal HE had, compared to healthy controls, increased latencies, decreased speed of voluntary and reflex saccads, more errors in anti-saccads, more anticipations saccads and more difficulties to fix the target.

Our hypothesis was that the use of the eye-tracker will enable the diagnosis of minimal HE by studying the characteristics of saccads and anti-saccads.

Since no gold-standard is available for the diagnosis of minimal HE, we will use the conclusion of an adjudication committee formed by 2 experts. Their clinical judgment will take into account the results of medical history, clinical examination, neuropsychological testing, PHES, Critical Flicker Frequency test (CFF), ammonemia levels, EEG and brain MRI with spectroscopy.

Gold standard definition: diagnostic of minimal HE as stated by adjudication committee composed of 2 experts. Each patient will be classified as : patient without EH (neither clinical or minimal) and patient with EHM. The results of medical history, clinical examination, EEG results (triphasic waves, decreased frequency), ammonia level (above 50mcmol/L or not), neuropsychological testing encompassing PHES (below -4 or not) and CFF (below 39Hz or not), brain MRI with MR-spectroscopy (HE profile on MRS) will be aggregated to obtain their adjudication. All the tests will be performed by trained personal aware of the evaluation of cirrhotic patients with possible HE. The eye-tracking evaluation will be blinded to the conclusion of the adjudication committee (presence or absence of HE).

Since the data from the eye-tracker are quantitative, a ROC curve will be used to evaluate the diagnostic performance of each parameters measured by the study device (mainly, saccads latencies, voluntary and reflexes ones, and the percentage of errors in saccads, anti-saccads and voluntary anticipations).

The ability of each measure to diagnose minimal HE will be evaluated by the area under the ROC and its 95% confidence interval. Sensibility, specificity, positive and negative predictive values will be given for each possible cut-off with their 95% confidence interval. In order to optimize the diagnostic performance, the most discriminating values will be used to build a multivariate diagnostic model. To prevent overfitting frequently associated with "standard" logistic regression, the selection of variables of interest will be performed with the LASSO method. This method is valuable when the number of subjects are limited.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for EHM+ subjects:

* Age between 18 and 70 (inclusive)
* Cirrhosis
* Minimal hepatic encephalopathy
* Expression of non opposition

Eligibility criteria for EHM- subjects:

* Age between 18 and 70 (inclusive)
* Cirrhosis
* No hepatic encephalopathy (minimal or clinical)
* Paired with EHM+ subjects about age, gender, MELD score and cirrhosis etiology
* Expression of non opposition

Exclusion Criteria for all subjects:

* Age older than 70
* MMS score < 24
* Clinical hepatic encephalopathy
* Cirrhosis etiology different from alcoholic, viral or metabolic one
* Intake of psychotropic drugs within 48h
* Alcohol intake > 30 g/j
* Heart, renal or respiratory failure
* Evolutive neurological diseases
* History of neurological diseases causing consequences
* Non corrected visuals disorders
* Oculomotor disorders from any etiology
* Highly-resistant bacteria carrier subjects
* Inability to put on the eye-tracker device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-10-17 (Estimated); Study Completion 2023-10-17 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance (evaluated with the area under the roc curve) associated with the measure of reflex saccads latencies for the diagnostic of minimal HE | one day
  The diagnostic performance of the measure of reflex saccads latencies will be evaluated by the area under the roc curve and its 95% confidence interval

SECONDARY OUTCOMES:
Area under the roc curve associated with the measure of reflex saccads speed for the diagnostic of minimal HE. | one day
  The diagnostic performance of the measure of reflex saccads speed will be evaluated by the area under the roc curve and its 95% confidence interval.
Association between reflex saccads speed and results of neuropsychological testings | one day
Area under the roc curve associated with the measure of reflex saccads gain for the diagnostic of minimal HE | one day
  The diagnostic performance of the measure of reflex saccads gain will be evaluated by the area under the roc curve and its 95% confidence interval.
Association between reflex saccads gain and results of neuropsychological testings | one day
Area under the roc curve associated with the measure of voluntary saccads latency for the diagnostic of minimal HE. | one day
  The diagnostic performance of the measure of voluntary saccads latency will be evaluated by the area under the roc curve and its 95% confidence interval.
Association between voluntary saccads latency and results of neuropsychological testings | one day
Area under the roc curve associated with the measure of voluntary saccads gain for the diagnostic of minimal HE. | one day
  The diagnostic performance of the measure of voluntary saccads gain will be evaluated by the area under the roc curve and its 95% confidence interval.
Association between voluntary saccads gain and results of neuropsychological testings | one day
Area under the roc curve associated with the measure of voluntary saccads anticipation for the diagnostic of minimal HE. | one day
  The diagnostic performance of the measure of voluntary saccads anticipation will be evaluated by the area under the roc curve and its 95% confidence interval.
Association between voluntary saccads anticipation and results of neuropsychological testings | one day
Area under the roc curve associated with the measure of percentage of errors in saccads for the diagnostic of minimal HE. | one day
  The diagnostic performance of the measure of percentage of errors in saccads will be evaluated by the area under the roc curve and its 95% confidence interval.
Association between percentage of errors in saccads and results of neuropsychological testings | one day
Area under the roc curve associated with the measure of percentage of errors in anti-saccads for the diagnostic of minimal HE | one day
  The diagnostic performance of the measure of percentage of errors in anti-saccads will be evaluated by the area under the roc curve and its 95% confidence interval.
Association between percentage of errors in anti-saccads and results of neuropsychological testings | one day

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas WEISS, MD, PhD, Principal Investigator — Pitié-Salpêtrière Hospital (AP-HP)
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France